CLINICAL TRIAL: NCT01681056
Title: Quality of Life and Psycho-Neuro-Endocrine-Immunology Pathway of Geriatric Patients: A Trial of Autosuggestion
Brief Title: Efficacy Study of Autosuggestion for Quality of Life of Geriatric Patients
Acronym: ESAQoGe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nina Kemala Sari, MD, Medical Doctor, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1134-1994
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Quality of Life for Geriatric Patients.
Keywords: autosuggestion; quality of life; geriatric; serum cortisol; Interferon gamma; interleukin-2; interleukin-6; neuroplasticity
MeSH Terms: interventions — Autosuggestion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autosuggestion (Experimental)
  Interventions: Behavioral: Autosuggestion for 30 days
- Standard medical theraphy (No Intervention)

INTERVENTIONS:
Behavioral: Autosuggestion for 30 days
  Other Names: Self talk
  Arms: Autosuggestion

SUMMARY:
The objective is to analyze the efficacy of autosuggestion for geriatric patients's quality of life and its impact to psycho-neuro-endocrine-immune pathways. The primary outcome is quality of life.

The hypothesis of this study is that autosuggestion will increase geriatric patient's quality of life based on its impact to psycho-neuro-endocrine-immune pathways.

DETAILED DESCRIPTION:
Geriatric patients diagnosed with multipathology after getting information and signing informed consent will be included in this trial. Autosuggestion was created by patients according to their preferences, modified by researcher to accomplish autosuggestion principles, recorded in a tape to be heard by walkman daily for 30 days. Intervention and control groups received usual standard medical therapy.

Baseline data were collected within one week after admission. Then the subject will be followed up for 30 days. Primary outcome was quality of life measured by COOP chart, analyze using on treatment analysis. Secondary outcomes were serum cortisol, interleukin-2, interleukin-6, IFN-ϒ (Interferon gamma), and N Acetyl Aspartat/ creatine ratio in limbic and paralimbic system by Magnetic Resonance Spectroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 60 years old with multipathology, inpatients
* Not in steroid therapy
* Could communicate (Karnofsky score: 40% or Zubrod/WHO score: 3)
* Cooperative
* Willing to go through all of the research steps.

Exclusion Criteria:

* Stroke
* Multiple Sclerosis
* Brain Tumour
* Using Pace maker

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life | 30 days
  Measured by COOP chart

SECONDARY OUTCOMES:
Serum Cortisol (ng/mL) | 30 days
  Change from baseline in Serum Cortisol concentration (ng/mL) measured by Radioimmunoassay method at 08.00-09.00 am.
Interleukin-2 (pg/mL) | 30 days
  Change from baseline in Interleukin-2 concentration (pg/mL) measured by ELISA method at 08.00-09.00 am.
Interleukin-6 (pg/mL) | 30 days
  Change from baseline in Interleukin-6 concentration(pg/mL) measured by ELISA method at 08.00-09.00 am.
Interferon Gamma (pg/mL) | 30 days
  Change from baseline in Interferon Gamma concentration (pg/mL) measured by ELISA method at 08.00-09.00 am.
N Acetyl Aspartat/ creatine ratio in limbic and paralimbic system (amygdala, hippocampus, hypothalamus, temporal lobe, accumbens nuclei, prefrontal cortex) | 30 days
  Ratio change from baseline by Magnetic Resonance Spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Nina K Sari, MD, Principal Investigator — Indonesia University
Locations (1):
- Dr. Cipto Mangunkusumo Hospital, Jakarta, DKI Jakarta, Indonesia